CLINICAL TRIAL: NCT01564329
Title: The Use of CT Perfusion to Determine the Normalization Window Period in the Treatment of Advanced Primary Lung Adenocarcinoma With Endostar
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: sim-endo-201201
Record Dates: First submitted 2012-03-21; First posted 2012-03-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Advanced Primary Lung Adenocarcinoma
Keywords: endostar; CT Perfusion; Advanced Primary Lung Adenocarcinoma
MeSH Terms: interventions — endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- endostar2 (Experimental): CT Perfusion Imaging(CTPI) at D0, D21 of the first cycle、D6, D14 of the second cycle, measure blood flow ( BF ), blood volume ( BV ), mean transit time ( MTT ), start time ( TTS ), time to peak ( TTP ), Patlak blood volume ( pBV ), vascular permeability etc. before/after tumor tissue treatment.
  Interventions: Drug: endostar
- endostar1 (Experimental): CT Perfusion Imaging(CTPI) at D0，D6, D14, D21 of the first period, measure blood flow ( BF ), blood volume ( BV ), mean transit time ( MTT ), start time ( TTS ), time to peak ( TTP ), Patlak blood volume ( pBV ), vascular permeability etc. before/after tumor tissue treatment.
  Interventions: Drug: endostar

INTERVENTIONS:
Drug: endostar — Endostar TM 7.5mg/m2,intravenous drip, Day 1to Day 10;Pemetrexed 500mg/m2, intravenous drip, Day 6; Carboplatin AUC=5,intravenous drip, Day 6; 21 days as a cycle, 4 cycles in all.

SUMMARY:
To evaluate the change of blood perfusion before/after the use of Endostar, discuss the time sequence of Endostar TM in treating advanced lung adenocarcinoma in normalization window period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically newly diagnosed as unresectable and metastasis advanced lung adenocarcinoma(Stage IV, Seventh Edition of the UICC/AJCC Classification for Lung Cancer).
* At least one measurable objective tumor lesion, spiral CT or PET-CT examination: the shortest diameter ≥2cm，and no obvious necrosis
* Life expectancy ≥12weeks
* Patients receive palliative radiotherapy for bone's pain relief; patients receive radiotherapy for brain metastasis、patients after brain transfer operation or radiation therapy are allowed to enter the research.
* 18≤Patients'age <70 years.
* Electrocolonogram (ECOG) Score:0-1.
* Granulocyte count ≥ 2.0×109/L, platelet count ≥ 100×109/L.
* Serum bilirubin within the normal range.
* Aspartate aminotransferase ( AST ), Alanine aminotransferase ( ALT ) within the normal range(if the patients is diagonosed as liver metastasis,his/her AST/ALT should not surpass 1.5 times of the normal range ).
* Serum creatinine within the normal range and creatinine clearance rate ≥60ml/min
* Compliance with research requirements and be able to follow up.
* Within 72 hours before the treatment, all women pregnant with pregnant possibility should undergo pregnancy test and get negative results.
* Patients with fertility ability should take effective contraceptive techniques.
* Sign informed consent of this clinic trial.

Exclusion Criteria:

* Lung adenocarcinoma patients who received systemic chemotherapy/thoracic radiotherapy/targeted therapy
* Received resection, cutting or aspiration within seven days
* Any unstable systemic diseases (including peptic ulcer、active infection、grade4 hypertension、unstable angina、congestive heart failure、liver, metabolic disorders or fracture、unhealing wound )
* Chronic kidney disease history(including chronic nephritis, nephrotic syndrome, Obstruction of urinary tract etc. caused by Urinary calculus)
* have to use anticoagulant drugs at the same time
* patients with obvious coagulation disorders、active bleeding and bleeding tendency
* Any other malignancies (complete cure of cervical carcinoma in situ/basal cell carcinoma/squamous cell carcinoma are excluded )happened within 5 years.
* Signifinant weight loss, weight lost during the 6 weeks more than or equal to 10%
* Patients who take bone metastasis as the only observing index
* Allergic to escherichia coli preparation
* Used Endostar before
* Lactating women
* Contraindications written on Pemetrexed、Carboplatin、Dexamethasone instructions
* Allergic to radiographic contrast agents
* In the middle or planning to attend other clinic trails

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-04 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
the change of blood perfusion before/after the use of Endostar | per 3 weeks

SECONDARY OUTCOMES:
tumor to progress | 6 months
  tumor to progress
clinical benefit rate | per 6 weeks
Adverse Drug Reaction | per 1 day
  NCI-CTCAE V3.0

CONTACTS AND LOCATIONS:
Locations (1):
- The Department of Thoracic Oncology in West China Hospital of Sichuan University, Chengdu, Sichuan, China